CLINICAL TRIAL: NCT00428519
Title: A Phase Ib, Randomized, Placebo Controlled, Double Blind Study to Determine the Safety, Viral Suppression, Pharmacokinetics and Immune Modulatory Effects of Treatment With Aprepitant (Emend®) in HIV Infected Individuals
Brief Title: Effects of Treatment With Aprepitant (Emend®) in HIV Infected Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 75558; U01MH090325 (NIH)
Record Dates: First submitted 2007-01-26; First posted 2007-01-30 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: HIV Infections
Keywords: HIV infection; Neurokinin-1 receptor antagonist; CCR5 expression; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Active Comparator)
  Interventions: Drug: Aprepitant
- 3 (Active Comparator)
  Interventions: Drug: Aprepitant

INTERVENTIONS:
Drug: Placebo — Placebo for 14 days
  Arms: 1
Drug: Aprepitant — Aprepitant at a dose of 125 mg daily for 14 days
  Arms: 2
Drug: Aprepitant — Aprepitant at a dose of 250 mg daily for 14 days
  Arms: 3

SUMMARY:
The investigators' in vitro data suggest that Neurokinin-1 receptor antagonists like aprepitant will decrease the expression of CCR5, an essential co-receptor in the life cycle of HIV, in the surface of macrophages and lymphocytes to levels at least similar to those observed in patients heterozygous for the CCR5 32 mutation. Together with a direct potential antiviral effect this could alter disease progression in patients with HIV infection.

The investigators' hypothesis is that aprepitant is safe, tolerable and has antiviral activity in HIV infected individuals.

This is randomized, placebo controlled, double blind study to determine the safety and antiviral activity of aprepitant by comparing the change in HIV RNA viral load after 2 weeks of aprepitant monotherapy.

27 HIV infected males and females ≥ 18 years old who have early infection with CD4 cell counts ≥ 350 cells/mm3. Subjects will be randomized 1:1:1 to receive two different doses of aprepitant (Emend®) or placebo.

DETAILED DESCRIPTION:
DESIGN

Randomized, placebo controlled, double blind study to determine the safety and antiviral activity of aprepitant by comparing the change in HIV RNA viral load after 2 weeks of aprepitant monotherapy.

DURATION

42 days.

SAMPLE SIZE and POPULATION

27 HIV infected males and females ≥ 18 years old who have early infection with CD4 cell counts ≥ 350 cells/mm3.

REGIMEN

Subjects will be randomized 1:1:1 to receive two different doses of aprepitant (Emend®) or placebo.

* Arm A: Aprepitant placebo
* Arm B: Aprepitant 125 mg QD
* Arm C: Aprepitant 250 mg QD

HYPOTHESIS AND STUDY OBJECTIVES

* Hypothesis : Aprepitant is safe, tolerable, and has antiviral activity in HIV infected individuals.
* Primary Objectives:

  * To assess the safety and tolerability of aprepitant for 2 weeks at two different doses.
  * To assess the response of plasma HIV-1 RNA to two different doses of aprepitant compared with baseline.
* Secondary Objectives:

  * To investigate the course and duration of antiretroviral response to 2 different doses of aprepitant given over a 14-day period.
  * To evaluate the dose-response and pharmacokinetic and pharmacodynamic relationship between viral RNA change and aprepitant plasma levels.
  * To evaluate aprepitant effects on CD4+ and CD8+ T-cell counts, circulating SP levels, natural killer cell number and function and CCR5 expression in peripheral PBMCs.
  * To evaluate the effects of aprepitant in the viral tropism and envelope sequence of the main HIV-1 population of the participants.
  * To assess viral drug susceptibility in conjunction with baseline coreceptor tropism phenotype and changes in coreceptor phenotype after the exposure to aprepitant.
  * To evaluate aprepitant effects on fasting plasma glucose, insulin, HDL, free fatty acids, and triglyceride concentrations after 14 days of treatment.
  * To provide preliminary description of any change from baseline in sleep quality, anxious mood, depressed mood and neurocognitive measures after 2 weeks of aprepitant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection, as documented by any licensed ELISA test kit and confirmed by Western blot at any time prior to study entry. HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test.
2. CD4+ cell count ≥ 350/mm3 obtained within 90 days prior to study entry and performed at any CLIA-certified laboratory.
3. Plasma HIV-1 RNA of ≥ 2000 copies/mL as measured by any standard assay (the Roche UltraSensitive HIV-1 Monitor assay (Roche Molecular Systems), or Version 3 bDNA assay or other) and performed within 90 days prior to study entry by any laboratory that is CLIA-certified (or its equivalent) for the assay.
4. CCR5 tropic virus exclusively as determined by the Monogram tropism assay (PhenoSense Entry™).
5. Laboratory values obtained within 30 days prior to study entry, as follows:

   * Absolute neutrophil count (ANC) greater than 750/mm3
   * Hemoglobin greater than 10.0 g/dL
   * Platelet count greater than 100,000/mm3
   * Creatinine less than 2 x ULN (fasting)
   * AST (SGOT), ALT (SGPT), and alkaline phosphatase less than 2 x ULN
   * Total bilirubin less than 2.5 x ULN
   * Albumin greater than 3 g/dL
   * Serum lipase less than 1.5 x ULN
6. Female subjects of reproductive potential must have a negative spot urine pregnancy test result (with a sensitivity of at least 50 mIU/mL) performed at entry, prior to starting initial study treatment.
7. All subjects must agree not to participate in a conception process while on study drug and for 30 days after stopping the medication.

   If participating in sexual activity that could lead to pregnancy, the female study subject must use at least one of the forms of contraception listed below while receiving the protocol-specified medication and for 30 days after stopping the medication:
   * Condoms (male or female) with or without a spermicidal agent
   * Diaphragm or cervical cap with spermicide
   * IUD

   Female subjects, who are not of reproductive potential defined as women who have been post-menopausal for at least 24 consecutive months, or women who have undergone surgical sterilization, (e.g. hysterectomy, bilateral oophorectomy, or salpingotomy) are eligible without requiring the use of contraception. Subject reported history is acceptable for documentation of sterilization, other contraceptive methods, menopause and a child's reproductive potential.
8. Karnofsky performance score greater than 80 within 30 days prior to study entry.
9. Men and women greater than 18 years of age.
10. Ability and willingness of subject or legal guardian/representative to give written informed consent.
11. Willing to return for a follow-up visit on day 42.
12. Subjects taking any precautionary concomitant medications must be on stable doses for > 8 weeks prior to study entry and have no plans to change medications or doses for the duration of the study.

Exclusion Criteria:

1. Receipt of antiretroviral treatment within the 16 weeks prior to study entry or intent to initiate antiretroviral therapy within 60 days after entry.
2. Diabetes requiring treatment with oral hypoglycemics or insulin therapy.
3. Pregnancy within 90 days prior to study entry.
4. Breast-feeding.
5. Use of drugs that are inhibitors or inducers of metabolism by the cytochrome P450 CYP3A4 or CYP2C9 (such as warfarin and phenytoin) within 7 days of study entry.
6. Use of systemic corticosteroids or hormonal agents within 90 days prior to study entry.
7. Use of any immunomodulator, HIV vaccines, or investigational therapy within 90 days prior to study entry.
8. Any vaccination within 30 days prior to study entry.
9. Use of systemic cytotoxic chemotherapy within 90 days prior to study entry.
10. History of allergy to aprepitant or its formulations.
11. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
12. History of chronic active hepatitis B or C infection or severe hepatic dysfunction (Child-Plug score > 9) regardless of etiology.
13. Serious illness requiring systemic treatment and/or hospitalization until subject either completes therapy or is clinically stable on therapy, in the opinion of the investigator, for at least 14 days prior to study entry.
14. Weight < 40 kg or 88 lbs within 90 days prior to study entry.
15. History of severe psychiatric comorbidities, such as depression, schizophrenia, mania, psychosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Virologic: Change in log10 HIV-1 RNA from baseline to Day 14 | 14 days
Safety: Incidence of Grade 2, 3, and 4 adverse events | 42 days

SECONDARY OUTCOMES:
Pharmacokinetic | 14 days
Immunologic | 14 days
Neurologic | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Tebas, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Clinical Trials Unit. University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Lai JP, Ho WZ, Zhan GX, Yi Y, Collman RG, Douglas SD. Substance P antagonist (CP-96,345) inhibits HIV-1 replication in human mononuclear phagocytes. Proc Natl Acad Sci U S A. 2001 Mar 27;98(7):3970-5. doi: 10.1073/pnas.071052298. PMID 11274418
- [Background] Lai JP, Ho WZ, Kilpatrick LE, Wang X, Tuluc F, Korchak HM, Douglas SD. Full-length and truncated neurokinin-1 receptor expression and function during monocyte/macrophage differentiation. Proc Natl Acad Sci U S A. 2006 May 16;103(20):7771-6. doi: 10.1073/pnas.0602563103. Epub 2006 May 4. PMID 16675550
- [Background] Ho WZ, Evans DL, Douglas SD. Substance P and Human Immunodeficiency Virus Infection: Psychoneuroimmunology. CNS Spectr. 2002 Dec;7(12):867-874. doi: 10.1017/s1092852900022483. PMID 12766696
- [Background] Ho WZ, Lai JP, Li Y, Douglas SD. HIV enhances substance P expression in human immune cells. FASEB J. 2002 Apr;16(6):616-8. doi: 10.1096/fj.01-0655fje. PMID 11919172
- [Background] Li Y, Douglas SD, Song L, Sun S, Ho WZ. Substance P enhances HIV-1 replication in latently infected human immune cells. J Neuroimmunol. 2001 Dec 3;121(1-2):67-75. doi: 10.1016/s0165-5728(01)00439-8. PMID 11730941
- [Result] Tebas P, Tuluc F, Barrett JS, Wagner W, Kim D, Zhao H, Gonin R, Korelitz J, Douglas SD. A randomized, placebo controlled, double masked phase IB study evaluating the safety and antiviral activity of aprepitant, a neurokinin-1 receptor antagonist in HIV-1 infected adults. PLoS One. 2011;6(9):e24180. doi: 10.1371/journal.pone.0024180. Epub 2011 Sep 8. PMID 21931661
- [Result] Tebas P, Spitsin S, Barrett JS, Tuluc F, Elci O, Korelitz JJ, Wagner W, Winters A, Kim D, Catalano R, Evans DL, Douglas SD. Reduction of soluble CD163, substance P, programmed death 1 and inflammatory markers: phase 1B trial of aprepitant in HIV-1-infected adults. AIDS. 2015 May 15;29(8):931-9. doi: 10.1097/QAD.0000000000000638. PMID 25915168